CLINICAL TRIAL: NCT04846712
Title: Interest of Ultrasound in the Diagnosis of Severity of Lateral Ankle Sprain
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN1382021/CHUSTE
Record Dates: First submitted 2021-04-13; First posted 2021-04-15 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Ankle Sprains
Keywords: Ankle; sprain; diagnosis; ultrasound; MRI
MeSH Terms: conditions — Ankle Injuries; Sprains and Strains; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with a first ankle sprain: 50 patients with a first ankle sprain will be included. Data will be collected of medical record.
  Interventions: Other: Collect data of medical record

INTERVENTIONS:
Other: Collect data of medical record — Collect data of medical record: initial physical examination, ultrasound (US), Magnetic Resonance Imaging (MRI), physical examination at 30 days, physical examination at 3 months, physical examination at 6 months and final examination at 12 months.

SUMMARY:
Ankle sprain is a frequent and widely trivialized trauma. Misdiagnosed or poorly treated, it can recur and thus develop into chronic ankle instability. It can be associated with complications which, if not detected early, can lead to long-term sequelae.

DETAILED DESCRIPTION:
The hypothesis of this study is that ultrasound can better characterize the severity stages of the sprain and can diagnose complications that may have gone unnoticed on physical examination.

Patients were assessed clinically: demographics, history, clinical examination, functional scores. An ultrasound and an MRI were done during the first month to check for complications. The main objective is to assess the value of ultrasound in the diagnosis of the severity of the lateral ankle sprain. The secondary objective is to compare an ultrasound assessment of severity with a clinical assessment and Magnetic Resonance Imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* First ankle sprain with sport or work disability

Exclusion Criteria:

* Patient with fractures, dislocation or hyperlaxity
* Previous ankle sprain

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with a first ankle sprain will be included.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Severity score by ultrasound (US) assesment | Day: 14 after Ankle Sprain.
  Collected in medical record.
  This system utilises a classification that is based on injury severity related to the amount of tissue damage and associated functional loss. It categorises muscle injuries into three grades, ranging from grade 1 with no appreciable tissue tear, grade 2 with tissue damage and reduced strength of the musculotendinous unit and grade 3 with complete tear of musculotendinous unit and complete loss of function

SECONDARY OUTCOMES:
Severity score by Magnetic Resonance Imaging (MRI) assesment | Day: 14 after Ankle Sprain.
  Collected in medical record.
  This system utilises a classification that is based on injury severity related to the amount of tissue damage and associated functional loss. It categorises muscle injuries into three grades, ranging from grade 1 with no appreciable tissue tear, grade 2 with tissue damage and reduced strength of the musculotendinous unit and grade 3 with complete tear of musculotendinous unit and complete loss of function
Severity score by radiologist assesment | Day: 30, 90, 180, 365 after Ankle Sprain.
  Collected in medical record.
  Empirical score : low, mild, severe

CONTACTS AND LOCATIONS:
Overall Officials: Thomas NERI, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No